CLINICAL TRIAL: NCT06801821
Title: Evaluation of Stigma Toward Patients With Alopecia Areata, Atopic Dermatitis, Vitiligo, and Psoriasis
Acronym: STIGMADERM
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7261
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis (PsO); Vitiligo Vulgaris; Atopic Dermatitis; Areata Alopecia
MeSH Terms: conditions — Psoriasis; Vitiligo; Dermatitis, Atopic; Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective:

The primary objective is to evaluate in the general population the difference between emotional reactions associated with facial involvement by four major dermatologic diseases: psoriasis, atopic dermatitis, vitiligo, and alopecia areata.

* Compare the social distance and stereotyping by the general population toward individuals with facial involvement by: psoriasis, atopic dermatitis, vitiligo, and alopecia areata.
* Evaluate demographic factors that describe a greater tendency toward stigmatization.

DETAILED DESCRIPTION:
Basic demographic characteristics (Gender, Age, Employment status, Education level) will be recorded for each patient.

Participants will be asked to observe images depicting faces of individuals with atopic dermatitis, alopecia areata, vitiligo, and psoriasis (generated through artificial intelligence systems). They will be asked to select the individual from those shown that generates the most compassion/pity, disgust, blame/disapproval/disdain, and curiosity for them, analyzing the same emotional responses investigated in a study on stigma toward psoriasis patients.

In addition, each participant will be given a 14-question questionnaire on stigma (analyzing social distance and stereotyping) toward one of the four diseases under investigation (psoriasis, atopic dermatitis, vitiligo, or alopecia areata), selected randomly. For each question, responses will be expressed from 1 to 5, on a Likert scale, with lower scores indicating greater stigma. (Total score between 14 and 70)

ELIGIBILITY:
Inclusion Criteria:

* -Patients aged>18 years, both sexes;
* Signature of written informed consent;

Exclusion Criteria:

* Patients diagnosed with psoriasis, atopic dermatitis, vitiligo or alopecia areata.
* Patients with first-degree relatives with psoriasis, atopic dermatitis, vitiligo or alopecia areata
* Those who for professional or personal reasons have direct knowledge of the diseases in question.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The intent of this observational study is primarily descriptive. It is estimated to be able to enroll 400 subjects adhering to the inclusion and exclusion criteria under treatment at the dermatology laboratory. Patients will be enrolled consecutively from 01-02-2025 to 01-02-2026. The 400 patients will answer initial questions about the emotional reactions induced by the 4 diseases and SYNOPSIS_STYGMADERM Study Version 1.0 on 03.10.24 Page 4 of 6 then will answer the questionnaire on stigma toward only one of the 4 dermatologic diseases under study (100 will answer the questionnaire on atopic dermatitis, 100 on alopecia areata, 100 on vitiligo, and 100 on psoriasis).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
primary endopoint | 12 months
  Compare the percentage of patients associating the 4 different emotional reactions analyzed (compassion/pity, disgust, blame/disapproval/dislike, and curiosity) with each dermatologic condition under study.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Caldarola, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Dermatologia, Roma, Italia, Italy